CLINICAL TRIAL: NCT01937377
Title: GLORIA-AF: Global Registry on Long-Term Oral Anti-thrombotic Treatment In Patients With Atrial Fibrillation (Phase II/III-India and Switzerland)
Brief Title: GLORIA-AF Registry Program (Phase II/III)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.171
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Stroke; Atrial Fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
In this part of the Registry Program patients with non-valvular atrial fibrillation (AF) at risk for stroke are enrolled to characterize the target population and to collect real world data on important outcome events.

For administrative purposes the study is divided into three protocol numbers: 1160.129 for all non-EU (European Union) and non-EEA (European Economic Area) countries, 1160.136 for EU and EEA countries and 1160.171 for Switzerland. The total number of patients enrolled in three protocols is estimated to be 48,000 patients, and all these patients will be included in the data analysis for study 1160.129.

ELIGIBILITY:
Inclusion criteria:

1) Patients newly diagnosed with non-valvular atrial fibrillation (NVAF) at risk for stroke.

Further inclusion criteria apply

Exclusion criteria:

1. Presence of any mechanical heart valve, or valve disease that is expected to require valve replacement intervention;
2. Patients who have received more than 60 days of vitamin K antagonist (VKA) treatment in their lifetime;
3. AF with a generally reversible cause;
4. Patients with a medical condition other than atrial fibrillation for which chronic use of an oral anticoagulant (for example, a VKA) is indicated.

Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with non-valvular AF
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-09-02 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Stroke (hemorrhagic and ischemic, uncertain classification) | up to 3 years
  The analysis of the outcome measure is included in study 1160.129
Systemic embolism | up to 3 years
  The analysis of the outcome measure is included in study 1160.129
Pulmonary embolism | up to 3 years
  The analysis of the outcome measure is included in study 1160.129
Myocardial infarction | up to 3 years
  The analysis of the outcome measure is included in study 1160.129
Life-threatening bleeding events | up to 3 years
  The analysis of the outcome measure is included in study 1160.129
All cause death | up to 3 years
  The analysis of the outcome measure is included in study 1160.129
Vascular death | up to 3 years
  The analysis of the outcome measure is included in study 1160.129
Major bleeding events (including life-threatening bleeding events) | up to 3 years
  The analysis of the outcome measure is included in study 1160.129
composite endpoint: Stroke, systemic embolism, myocardial infarction, life-threatening bleeding events and vascular death | up to 3 years
  The analysis of the outcome measure is included in study 1160.129
composite endpoint: Stroke, systemic embolism, myocardial infarction and vascular death (vascular composite endpoint) | up to 3 years
  The analysis of the outcome measure is included in study 1160.129
Transient Ischemic Attack (TIA) | up to 3 years
  The analysis of the outcome measure is included in study 1160.129

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- Switzerland (5):
  - University Hospital Basel, Basel
  - CHUV - Centre hospitalier universitaire vaudois, Lausanne
  - Cardiocentro Ticino, Lugano
  - Kantonsspital St.Gallen, Sankt Gallen
  - Arzte Zentrum Eigerpark, Urtenen-Schonbuhl, Schönbühl

REFERENCES:
- [Derived] Joddrell M, El-Bouri W, Harrison SL, Huisman MV, Lip GYH, Zheng Y; GLORIA-AFinvestigators. Machine learning for outcome prediction in patients with non-valvular atrial fibrillation from the GLORIA-AF registry. Sci Rep. 2024 Nov 7;14(1):27088. doi: 10.1038/s41598-024-78120-z. PMID 39511367
- [Derived] Romiti GF, Corica B, Proietti M, Mei DA, Frydenlund J, Bisson A, Boriani G, Olshansky B, Chan YH, Huisman MV, Chao TF, Lip GYH; GLORIA-AF Investigators. Patterns of oral anticoagulant use and outcomes in Asian patients with atrial fibrillation: a post-hoc analysis from the GLORIA-AF Registry. EClinicalMedicine. 2023 Aug 25;63:102039. doi: 10.1016/j.eclinm.2023.102039. eCollection 2023 Sep. PMID 37753446
- [Derived] Ding WY, Fawzy AM, Romiti GF, Proietti M, Pastori D, Huisman MV, Lip GYH; GLORIA-AF Investigators. Validating the predictive ability of the 2MACE score for major adverse cardiovascular events in patients with atrial fibrillation: results from phase II/III of the GLORIA-AF registry. J Thromb Thrombolysis. 2024 Jan;57(1):39-49. doi: 10.1007/s11239-023-02866-y. Epub 2023 Aug 11. PMID 37566295
- [Derived] Ding WY, Lane DA, Gupta D, Huisman MV, Lip GYH; GLORIA-AF Investigators. Incidence and Risk Factors for Residual Adverse Events Despite Anticoagulation in Atrial Fibrillation: Results From Phase II/III of the GLORIA-AF Registry. J Am Heart Assoc. 2022 Aug 2;11(15):e026410. doi: 10.1161/JAHA.122.026410. Epub 2022 Jul 25. PMID 35876418
- [Derived] Ding WY, Calvert P, Gupta D, Huisman MV, Lip GYH; GLORIA-AF Investigators. Impact of early ablation of atrial fibrillation on long-term outcomes: results from phase II/III of the GLORIA-AF registry. Clin Res Cardiol. 2022 Sep;111(9):1057-1068. doi: 10.1007/s00392-022-02022-1. Epub 2022 Apr 29. PMID 35488127
- [Derived] Azar RR, Ragy HI, Kozan O, El Khuri M, Bazergani N, Marler S, Teutsch C, Ibrahim M, Lip GYH, Huisman MV. Antithrombotic treatment pattern in newly diagnosed atrial fibrillation patients and 2-year follow-up results for dabigatran-treated patients in the Africa/Middle-East Region: Phase II results from the GLORIA-AF registry program. Int J Cardiol Heart Vasc. 2021 Apr 10;34:100763. doi: 10.1016/j.ijcha.2021.100763. eCollection 2021 Jun. PMID 33912651
- [Derived] Ntaios G, Huisman MV, Diener HC, Halperin JL, Teutsch C, Marler S, Gurusamy VK, Thompson M, Lip GYH, Olshansky B; GLORIA-AF Investigators. Anticoagulant selection in relation to the SAMe-TT2R2 score in patients with atrial fibrillation: The GLORIA-AF registry. Hellenic J Cardiol. 2021 Mar-Apr;62(2):152-157. doi: 10.1016/j.hjc.2020.11.009. Epub 2020 Dec 15. PMID 33338644
- [Derived] Huisman MV, Rothman KJ, Paquette M, Teutsch C, Diener HC, Dubner SJ, Halperin JL, Ma CS, Zint K, Elsaesser A, Lu S, Bartels DB, Lip GYH; GLORIA-AF Investigators. Two-year follow-up of patients treated with dabigatran for stroke prevention in atrial fibrillation: Global Registry on Long-Term Antithrombotic Treatment in Patients with Atrial Fibrillation (GLORIA-AF) registry. Am Heart J. 2018 Apr;198:55-63. doi: 10.1016/j.ahj.2017.08.018. Epub 2017 Aug 31. PMID 29653649
- See also: Results of this study are submitted together with study 1160.129 — https://clinicaltrials.gov/ct2/show/results/NCT01468701?term=1160.129&draw=2&rank=1